CLINICAL TRIAL: NCT03254381
Title: The Effect of Resistance Training on Cognitive Function and Brain Health in Older Adults At-risk for Diabetes: A Feasibility Pilot Study
Brief Title: The Effect of Exercise on Cognition in Older Adults At-risk for Diabetes: A Feasibility Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Lindsay Nagamatsu, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109379
Record Dates: First submitted 2017-08-03; First posted 2017-08-18 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Cognitive Impairment
Keywords: cognitive assessment; cognitive function; community dwelling older people; pre-diabetes; randomized control trial; exercise; pilot study; feasibility study
MeSH Terms: conditions — Cognitive Dysfunction; Glucose Intolerance; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Training (Experimental): Participants will use programmable weight machines along with free weights to target primary muscle groups. In addition, they will complete mini-squats, mini-lunges, and lunge walks. Participants will complete two sets of 6-8 reps. Training stimulus will be increased using the 7RM method - when 2 sets of 6-8 reps are completed with proper form and without discomfort. Investigators will record the number of sets completed and the load lifted for each exercise for each participant at every class.
  Interventions: Behavioral: Resistance Training
- Balance and Tone Training (Control) (Experimental): Exercises will include stretching exercises, range of motion exercises, basic core-strength exercises, balance exercises, and relaxation techniques. Only bodyweight will be applied (i.e., no additional loading). This group controls for confounding variables such as physical training received by traveling to the training centres, social interaction, and changes in lifestyle secondary to study participation.
  Interventions: Behavioral: Balance and Tone Training

INTERVENTIONS:
Behavioral: Resistance Training — Six months of thrice-weekly resistance training that will gradually progress in intensity. Each training session will be 60 minutes (10 minutes of warm-up, 40 minutes of training, and 10 minutes of cool-down). Classes will be group classes, with up to five participants in each.
  Arms: Resistance Training
Behavioral: Balance and Tone Training — Six months of thrice-weekly stretching and relaxation exercises. Each session will be 60 minutes. Classes will be group classes, with up to five participants in each.
  Arms: Balance and Tone Training (Control)

SUMMARY:
Older adults with type 2 diabetes experience cognitive decline and are at higher risk for developing dementia. Consequently, older adults at-risk for developing type 2 diabetes (based on body mass, glucose levels) are at higher risk for cognitive decline, and intervening at this point may prevent or delay the onset of such decline. One promising lifestyle intervention that has been shown to improve cognitive function in other populations is exercise. However, before investigators can examine whether exercise will improve cognitive function and brain health (structure and function) in this at-risk population, a feasibility pilot study is needed to determine whether a larger-scale trial would be viable.

DETAILED DESCRIPTION:
Investigators will conduct a six-month randomized control trial (RCT) exercise intervention. Thirty older adults (aged 60-80) at-risk for diabetes will be randomly assigned into one of two groups: 1) Resistance training, or 2) Balance and Tone training (control). All participants will engage in three one-hour exercise classes per week. Once a month, a neutral assessor will visit the classes to evaluate the quality of the classes for participants. Assessments will be made at baseline, midpoint (three months) and trial completion (six months), and will include cognitive testing, health questionnaires, physical testing, and magnetic resonance imaging (MRI; to assess structural and functional brain changes). Throughout the study, investigators will examine data for trends in successful recruitment strategies and rates of recruitment and adherence to inform future clinical trials in this population. Research assistants (n = 30) in the study will complete an anonymous feedback survey upon completion of their volunteer term, to assist in improving the study for future participants and volunteers.

ELIGIBILITY:
Inclusion Criteria:

1) be community-dwelling 2) be aged 60-80 years 3) be "at-risk" for diabetes, where they have one of the following: i) blood glucose level of 6.1-7 mmol/L, ii) BMI > 25, or iii) score > 21 on the CANRISK diabetes questionnaire 4) score > 24/30 on MMSE 5) score > 6/8 on Lawton and Brody's Independent Activities of Daily Living (IADL) scale 6) have visual acuity of at least 20/40, with or without corrective lenses 7) speak and understand English fluently 8) complete the Physical Activity Readiness Questionnaire (PAR-Q) 9) obtain physician's clearance to start a supervised exercise program

Exclusion Criteria:

1) have a current medical condition for which exercise is contraindicated 2) have participated regularly in resistance or aerobic training in the last 6 months 3) have been diagnosed with neurodegenerative disease (including dementia, Alzheimer's disease, or Parkinson's disease) 4) have experienced a vascular incident (e.g., stroke, myocardial infarction) 5) have been diagnosed with a psychiatric condition 6) have untreated depression 7) are currently on hormone replacement therapy 8) have clinically significant peripheral neuropathy or severe musculoskeletal or joint disease 9) are currently taking psychotropic medications 10) are unable to participate in MRI (have metal or electronic implants, or are claustrophobic)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited after 12 months | 12 months
Number of exercise classes attended at trial completion (6 months) | 6 months

SECONDARY OUTCOMES:
Change in cognitive function as measured by Alzheimer's Disease Assessment Scale - Cog - Plus (ADAS-Cog-Plus) | Baseline, 3 months, and 6 months
Change in hippocampal volume as measured via high resolution T1 images collected during MRI scanning in both 3T and 7T machines. | Baseline and 6 months
Change in hippocampal functional activation as measured during performance on associative memory task during fMRI scanning | Baseline and 6 months
  For this task, participants will be asked to encode and then recall items (face or places) and items in conjunction (faces matched with places)
Change in memory as measured by performance on associative memory task | Baseline, 3 months, and 6 months
Change in executive functions as measured by Stroop Test | Baseline, 3 months, and 6 months
Change in aerobic fitness as measured by six minute walk test | Baseline, 3 months, and 6 months
Change in mobility and balance as measured by Short Physical Performance Battery | Baseline, 3 months, and 6 months
Change in muscle strength as measured by one-repetition maximum test | Baseline, 3 months, and 6 months
Change in blood glucose levels as measured by finger prick glucose test | Baseline, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay S Nagamatsu, Principal Investigator — Western University
Locations (1):
- Community, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furlano JA, Nagamatsu LS. Feasibility of a 6-month pilot randomised controlled trial of resistance training on cognition and brain health in Canadian older adults at-risk for diabetes: study protocol. BMJ Open. 2019 Oct 3;9(10):e032047. doi: 10.1136/bmjopen-2019-032047. PMID 31585978